CLINICAL TRIAL: NCT03794778
Title: Evaluation of PEGylated Doxorubicin Hydrochloride Liposome Injection(Duomeisu®) Combined With Carboplatin Versus Paclitaxel Plus Carboplatin in the First-line Treatment of Epithelial Ovarian Cancer: A Randomized, Open, Multicenter Clinical Study
Brief Title: Evaluation of PLD Combined With Carboplatin Versus Paclitaxel Plus Carboplatin in the First-line Treatment of Epithelial Ovarian Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Principal Investigator, Xing Xie, Dean of Women's Hospital School Of Medicine Zhejiang University, Women's Hospital School Of Medicine Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180148
Record Dates: First submitted 2018-12-24; First posted 2019-01-07 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Efficacy and Safety
Keywords: PEGylated Doxorubicin Hydrochloride Liposome Injection; Duomeisu; First-line treatment; Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — liposomal doxorubicin; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): pegylated liposomal doxorubicin 30 mg/m2, i.v.,d1; carboplatin AUC 5,i.v.,d1; once every 21days, 3~6 cycles for early stage patients and 6 cycles for late stage.
  Interventions: Drug: pegylated liposomal doxorubicin; Drug: Carboplatin
- chemotherapy (Active Comparator): paclitaxel 175 mg/m2, i.v.,d1; carboplatin AUC 5, i.v.,d1; once every 21days, 3~6 cycles for early stage patients and 6 cycles for late stage.
  Interventions: Drug: paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin — PLD 30 mg/m2, i.v.,d1; once every 21days
  Other Names: duomeisu
  Arms: study group
Drug: paclitaxel — paclitaxel 175 mg/m2, i.v.,d1; once every 21days
  Other Names: zishanchun
  Arms: chemotherapy
Drug: Carboplatin — carboplatin AUC 5, i.v.,d1; once every 21days,
  Other Names: kabo

SUMMARY:
This is a randomized, multicenter, open, controlled Post-Marketing Study. 396 patients who were histopathology or exfoliated cell pathology of pleural and ascites confirmed with epithelial ovarian cancer/fallopian tube/peritoneal cancer were enrolled in this study. The subjects will be randomly assigned to one of the two treatment groups at a 1: 1 ratio, and the stratification factors included: chemotherapy type (adjuvant chemotherapy/neoadjuvant chemotherapy), residual disease after surgery (>1cm, <1cm, no primary surgery), stage (Ic, II, III or IV), pathological typing, Eastern Cooperative Oncology Group performance status (0 to 1 or 2), BRCA1/2 gene mutation.

DETAILED DESCRIPTION:
Subjects will receive one of two treatment regimens:

Group A: intravenous infusion of liposomal doxorubicin 30 mg/m2, d1; carboplatin AUC 5 (dosed according to the Calvert formula, with creatinine clearance estimated according to the Cockcroftformula), intravenous infusion, d1; once every 21days, 3~6 cycles for early stage patients and 6 cycles for late stage.

Group B: intravenous infusion of paclitaxel 175 mg/m2, d1; carboplatin AUC 5, intravenous infusion, d1; once every 21days, 3~6 cycles for early stage patients and 6 cycles for late stage. Treatment was initially administered for three cycles, and patients with stable or responding disease continued treatment for further a three cycles.

The main purpose is to evaluate the efficacy and safety of liposomal doxorubicin plus carboplatin in the first-line treatment of epithelial ovarian cancer. The primary endpoint is progression free survival (PFS), the secondary endpoints include overall survival (OS), objective response rate (ORR), disease control rate (DCR):CR+PR+SD, the incidence and severity of adverse reactions and health-related quality of life (HQL) assessment.

ELIGIBILITY:
Inclusion Criteria:

* 18-75years old;
* Histopathologically or exfoliated cell pathology of pleural and ascites confirmed with epithelial ovarian cancer/fallopian tube/peritoneal cancer;
* According to the International Federation of Obstetrics and Gynecology (FIGO), the stage is Ic-IV;
* Imaging assessment is based on the solid tumor efficacy evaluation standard (RECIST) version 1.1, lesions can be measured, or patients' CA125 assessed according to GCIG criteria;
* Neoadjuvant chemotherapy can be given to patients with excessive tumor volume or a wide range of lesions, who are not expected to achieve ideal cytoreductions before surgery;
* ECOG score ≤ 2;
* Expected survival time ≥ 3 months;
* LVEF ≥ 50%;
* Bone Marrow Function: ANC：≥1.5×109/L； PLT：≥100×109/L；Hb: ≥90g/L;
* Liver and renal function:Serum creatinine ≤ normal upper limit (ULN) 1.5times; aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤ULN 2.5times, or <ULN 5times in the presence of liver metastasis; total bilirubin (TBil) level≤ ULN 1.5 times, or ≤ ULN 2.5times if Gilbert's syndrome are present;
* The childbearing age subjects must agree to take effective contraceptive measures during the trial; the serum or urine pregnancy test must be negative, non-lactating;
* Signed the informed consent.

Exclusion Criteria:

* Patients with low-grade malignant potential ovarian tumors;
* Patients who had previously received chemotherapy or pelvic and abdominal radiotherapy;
* Patients planning to receive abdominal or pelvic chemotherapy;
* The New York Heart Association (NYHA) graded class II heart disease patients (including grade II) previous or current;
* Other malignant tumors have been found in the past 5 years,except for cured cervical carcinoma in situ, non melanoma of the skin;
* Uncontrolled systemic infection requiring anti-infective treatment;
* Allergies to chemotherapeutic drugs or their excipients or intolerant patients;
* Subjects with ≥2 grade peripheral neuropathy according to CTCAE V 4.03;
* Researchers think it is not suitable for enrolling.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or death from any cause, whichever occurred first, or last follow-up for patients alive without progression, assessed up to approximately 36 months.
  PFS is defined as the time from randomization to the first occurrence of PD, as determined by the investigator using RECIST v1.1, or death from any cause during the study, whichever occurs first.

SECONDARY OUTCOMES:
OS | From date of randomization until the date of death from any cause, or date of last follow-up for patients still alive, assessed up to 36 months
  overall survival
ORR | From date of randomization until PD or death from any cause, assessed up to 36 months.
  ORR is defined as the rate of CR or PR, as determined by IRC using RECIST v1.1 criteria among patients with at least one target lesion. Activity was also described in women with nontarget lesions only and in women without any tumor lesion but with elevated CA-125 levels before starting treatment.
DCR | From date of randomization until PD or death from any cause, assessed up to 36 months.
  DCR is defined as the rate of of CR, PR, or stable disease according to RECIST v1.1.
the incidence and severity of adverse reactions | A summary of adverse events of each cycle,from date of administration of drugs until 30 days after the last chemotherapy or progression,whichever came first,assessed up to 36 months.
  Evaluate the adverse reactions rate of drugs assessed by number and severity of adverse events in the treatment.
quality of life assessment | It will be assessed at baseline and before the administration of drugs at each first day of every two chemotherapy cycles, up to 6 cycles,each cycle is 21 days.
  according to the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C30 (QLQ-C30).The basic content of life quality assessment includes: physical health, mental health, social function, disease status and overall health perception.

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Hospital School Of Medicine Zhejiang University, Zhejiang, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No